CLINICAL TRIAL: NCT02272907
Title: Comparison of Leak Pressure in the Resected Gastric Specimen From Sleeve Gastrectomy With Different Reinforcement Techniques
Brief Title: Leak Pressure After Reinforcement in Gastric Specimens
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Barbara Cottage Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14-27r
Record Dates: First submitted 2014-10-15; First posted 2014-10-23 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Obesity
Keywords: Bariatric Surgery; Laparoscopy; Weight Loss Surgery; Staple Line Reinforcement
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Non-buttressed, non-imbricated oversewing (Experimental): Along the staple line, the surgical attending will oversew the length of the staple line using a 2-0 Vicryl suture in a continuous fashion.
  Interventions: Other: Injection of saline solution into specimen to test bursting pressure.
- Non-buttressed, imbricated suture line (Experimental): Along the staple line, the surgical attending will oversew the staple line using a 2-0 Vicryl suture in a continuous, imbricating fashion.
  Interventions: Other: Injection of saline solution into specimen to test bursting pressure.
- Buttressed stapling (Experimental): The specimen will be stapled utilizing the same stapling device, with Seamguard applied as a buttress. We will use the standard methodology to apply Seamguard as illustrated in the company's "Instructions for Use."
  Interventions: Other: Injection of saline solution into specimen to test bursting pressure.
- No reinforcement (Active Comparator): Data will be collected on staple lines without any reinforcement as a baseline for leak pressure.
  Interventions: Other: Injection of saline solution into specimen to test bursting pressure.

INTERVENTIONS:
Other: Injection of saline solution into specimen to test bursting pressure. — A 1 cm gastrotomy will be made with a purse-string suture placed around the defect. A fluid-instillation catheter will be inserted into the specimen via the gastrotomy. The purse-string suture will then be secured around the catheter. The catheter will be fenestrated with a flange to prevent leakage from the gastrotomy site. The catheter will be attached to a Biopac pressure-monitoring device to monitor pressure within the lumen of the specimen. The specimen will then be suspended in a water bath and methylene blue saline solution will be injected into the specimen to a pressure reading of 0. This will be time zero for our experiment. Methylene blue saline solution will then be injected steadily in incremental levels. During this process, the study team will observe for any obvious blue dye leaks at the staple line or drop in pressure on the monitor.

SUMMARY:
The investigators hypothesize that staple line reinforcement will result in a higher leak pressure than a non-reinforced staple line closure in the resected gastric specimens from laparoscopic sleeve gastrectomy. The primary endpoint of the study is leak pressure after various staple line treatments. The investigators will also analyze the most common site of specimen leak, association of stomach thickness to leak, association of stomach thickness to performance of the staple line techniques, and a cost analysis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the mechanical strength of various staple line reinforcement techniques using the resected portion of stomach in patients undergoing laparoscopic sleeve gastrectomy. The specimen will be collected at the time of surgery, the previous staple line will be excised, and a new staple line with one of the investigatory reinforcement procedures will be applied. The staple line techniques to be used in this study include non-buttressed and non-imbricated oversewing, non-buttressed and imbricated suture line, buttressed stapling, and no reinforcement (see protocol for description of each). The specimen will then be taken to the morgue where the experimental procedure will be performed within 6 hours of specimen procurement. The specimen will be attached to a catheter with a pressure monitor and blue dye will be instilled into the specimen until leakage is seen. The presence of leakage indicates failure of the staple line. Detailed measurements of all specimens will be performed as will leak pressure and location in the specimen where leak occurred. The specimen will then be turned over to pathology to undergo routine pathologic examination.

This experimental procedure has been used previously in published literature with animal samples, but never with human tissue. A possible reason for the lack of testing in the stomach staple line in patients after sleeve gastrectomy is that the technical aspects of bariatric surgery were developed using gastric bypass; a procedure where the stomach is divided but not excised.

The investigators hypothesize that the specimens treated with staple line buttressing material will fail at a higher pressure than those without reinforcement. The investigators will also explore the location of the failure to determine if there is a consistent site of weakness. Should this study yield consistent results, it would help determine a standard approach for staple line reinforcement after laparoscopic sleeve gastrectomy. Additionally, should the location of the leak be consistent, this information may help drive technical changes that could decrease leak rate, an infrequent but potentially devastating risk of this and other weight loss surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing laparoscopic sleeve gastrectomy

Exclusion Criteria:

* Undergoing a revisional procedure
* Subject whose specimens need clinical attention by pathology following resection (e.g. cancer biopsy)
* Steroid use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Bursting pressure | This will be measured within 6 hours of the specimen being resected from the patient.
  The primary outcome will be assessed by inflating the resected stomach specimen (after staple line reinforcement and placement of pressure monitor within specimen) with a methylene blue saline solution until a leak is observed or drop in pressure on the monitor.

SECONDARY OUTCOMES:
Most common leak site | This will be measured within 6 hours of the specimen being resected from the patient.
  The site of leak will be documented. This outcome will be observed by the individual testing the leak pressure of the specimen.